CLINICAL TRIAL: NCT00294866
Title: An Open Label, Multi-Center Study of the Effect of Paricalcitol on Markers of Inflammation in Patients With Stage 5 Chronic Kidney Disease on Hemodialysis.
Brief Title: Effect of Paricalcitol on Markers of Inflammation in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Mark Kaplan, M.D., Vice President of Clinical Research, Fresenius Medical Care North America
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2005002
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Kidney Failure
Keywords: End Stage Renal Disease; Inflammation
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Inflammation | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Receive Paricalcitol
  Interventions: Drug: Paricalcitol
- B (No Intervention): Paricalcitol on hold
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Patients randomized to either receive Paricalcitol or have it held. After 4 weeks they are switched to the opposite intervention.

SUMMARY:
Studies have shown that patients with ESRD on hemodialysis have high levels of inflammatory markers which may contribute to the high rates of cardiovascular disease and mortality seen in these patients. Vitamin D use in dialysis patients has been shown to have a survival benefit, with paricalcitol at advantage over calcitriol. Since there is some evidence for involvement of the vitamin D receptor in inflammation, this study is designed to look for an effect of paricalcitol on markers of inflammation in hemodialysis patients.

DETAILED DESCRIPTION:
Patients with ESRD have a high incidence of acute phase inflammation. Studies have shown that C-reactive Protein (CRP) and interleukin-6 (IL-6) are excellent biomarkers for inflammation, and high levels are predictive of cardiovascular morbidity and mortality in this population. Both uremia and the dialysis process itself contribute to this inflammatory state. It is our hypothesis that paricalcitol therapy decreases the biomarkers of inflammation which may have implications for future studies of morbidity and mortality in this population.

ELIGIBILITY:
Inclusion Criteria:

1. CKD and receiving hemodialysis for greater than or equal to 3 months
2. Age greater than or equal to 18 years
3. Medically stable
4. AVF or PTFE dialysis access
5. No acute inflammatory disease within 4 weeks prior to study
6. On an average dose of 3 - 7 mcg of paricalcitol three times per week for 4 weeks prior to the study
7. Two consecutive iPTH of 150-400 (biPTH 75 - 200) =/- 30% one week apart
8. Ca <10.2 mg/dL; PO4 <7.0
9. Kt/V greater than or equal to 1.2
10. On no other interventional drugs/devices in the past 30 days

Exclusion Criteria:

1. Currently receiving dialysis using a venous catheter access
2. Currently receiving high dose immunosuppressive therapy (greater than or equal to 10 mg prednisone)
3. Pregnancy
4. Hospitalization within the last 4 weeks. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome is a 20% change in IL-6 as a function of paricalcitol therapy. | 4 weeks

SECONDARY OUTCOMES:
Secondary Outcome is a significant change in markers of inflammation to include: | 4 weeks
CRP,TNFα, IL-1β, IL-8, IL-10, IL-12p70, PTH, Ca/P | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Kaplan, M.D., Principal Investigator — Fresenius Medical Care North America
Locations (6):
- United States (6):
  - Southwest Nephrology, Evergreen Park, Illinois
  - Nephrology Center, Kalamazoo, Michigan
  - Nephrology Associates P.A., West Orange, New Jersey
  - Delaware Valley Nephrology, Philadelphia, Pennsylvania
  - Nephrology Associates, PC, Nashville, Tennessee
  - Tyler Nephrology Associates, Tyler, Texas